CLINICAL TRIAL: NCT04145492
Title: The Impact of Vitamin K2 and Inactive Vitamin D Supplementation on Vascular Calcification in Pediatric Patients on Regular Hemodialysis
Brief Title: Effect of Vitamin K 2 on Vascular Calcification in Hemodialysis Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Maher Abd El Kader El Borolossy, lecturer of clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis and Vitamin K2
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Vitamin K 2; Cholecalciferol; Calcifediol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vitamin K2 group (Active Comparator): 15 patients will take 90 ug of vitamin K2 (MK-7) daily in addition to the standard therapy for 4 months.
  Interventions: Drug: Vitamin K2
- Cholecalciferol group (Active Comparator): 15 patients will take 10 ug of vitamin inactive vitamin D daily in addition to the standard therapy for 4 months.
  Interventions: Drug: Cholecalciferol (inactive vitamin D)
- Vitamin K2 and Cholecalciferol group (Active Comparator): 15 patients will take 90 ug of vitamin K2 (MK-7) in addition 10 ug of vitamin inactive vitamin D to daily in addition to the standard therapy for 4 months.
  Interventions: Drug: Cholecalciferol (inactive vitamin D); Drug: Vitamin K2 and Cholecalciferol
- Control group (No Intervention): 15 patients will take the standard therapy.

INTERVENTIONS:
Drug: Vitamin K2 — Patients will take 90 ug of vitamin K2
  Other Names: Group 1
  Arms: Vitamin K2 group
Drug: Cholecalciferol (inactive vitamin D) — Patients will take 10 ug of vitamin inactive vitamin D
  Other Names: Group 2
  Arms: Cholecalciferol group; Vitamin K2 and Cholecalciferol group
Drug: Vitamin K2 and Cholecalciferol — Patients will take 90 ug of vitamin K2 (MK-7) in addition 10 ug of vitamin inactive vitamin D
  Other Names: Group 3
  Arms: Vitamin K2 and Cholecalciferol group

SUMMARY:
The aim of this study is to assess the effect of supplementation of vitamin K2 (menaquinone, MK-7) and cholecalciferol (inactive vitamin D) on circulating levels of calcification regulators and to assess their safety in pediatric patients on regular hemodialysis patients.

DETAILED DESCRIPTION:
Vascular calcification occurs in more than half of chronic renal failure patients, which mainly appears in the large and medium size arteries [3, 4]. It seems that vas¬cular calcification is caused by dynamic imbal-ance of intravascular calcium and phosphorus. However, more and more studies pointed out that vascular calcification were related with local cell's function and biological characteris¬tics.

The aim of this study is to assess the effect of supplementation of vitamin K2 (menaquinone, MK-7) and cholecalciferol (inactive vitamin D) on circulating levels of calcification regulators and to assess their safety in pediatric patients on regular hemodialysis patients.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 6-18 years
* Patients on hemodialysis since 3 months or longer
* Hemodialysis frequency 3 times or more weekly

Exclusion criteria:

* Patients with life expectancy < 3 months
* Patients taking warfarin
* Patients with known intestinal malabsorption

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Uncarboxylated MGP | 4 months
  Measuring serum level of Uncarboxylated MGP as a marker for calcification
Uncarboxylated osteocalcin | 4 months
  Measuring serum level of Uncarboxylated osteocalcin as a marker for calcification

CONTACTS AND LOCATIONS:
Locations (1):
- Radwa Maher El Borolossy, Cairo, Egypt

REFERENCES:
- [Derived] El Borolossy R, El-Farsy MS. The impact of vitamin K2 and native vitamin D supplementation on vascular calcification in pediatric patients on regular hemodialysis. A randomized controlled trial. Eur J Clin Nutr. 2022 Jun;76(6):848-854. doi: 10.1038/s41430-021-01050-w. Epub 2021 Nov 29. PMID 34845313